CLINICAL TRIAL: NCT06676527
Title: An Observational Study of the Efficacy and Safety of Vorolanib in the Second-line Treatment of Patients With Unresectable or Metastatic Renal Cell Carcinoma
Brief Title: Vorolanib in the Second-line Treatment of Patients With Unresectable or Metastatic Renal Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Other Study IDs: 2024DZKY-074-02
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Female Urogenital Diseases; Male Urogenital Diseases; Urogenital Diseases; Kidney Diseases; Urologic Diseases; Carcinoma; Renal Cell Cancer; Carcinoma, Renal Cell; Antineoplastic Agents
Keywords: observational study; clear cell Renal Cell Carcinoma; TKIs
MeSH Terms: conditions — Neoplasms; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Female Urogenital Diseases; Male Urogenital Diseases; Urogenital Diseases; Kidney Diseases; Urologic Diseases; Carcinoma; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental cohort.: Subjects who progressed after first-line treatment and switched to second-line treatment regimens including vorolanib. The first-line treatment which patients received can be other tyrosine kinase inhibitors (TKIs) or TKIs combined with immunotherapy drugs. Provided vorolanib is contained in the second-line regimen, the patient then can be considered for inclusion in the study.
  Interventions: Other: Follow-up study of the treated cohort

INTERVENTIONS:
Other: Follow-up study of the treated cohort — For those patients who have reached the end point of the study, survival data during treatment with vorolanib is obtained for retrospective analysis. The patients who are still on treatment with vorolanib are followed up closely and survival data is obtained for prospective analysis. After summarizing the results of retrospective and prospective studies, relevant efficacy and safety conclusions will be drawn.

SUMMARY:
This is a multicenter real world study (RWS) initiated by the investigator. Eligible patients will be selected for treatment with second-line treatment including vorolanib and followed up. The real survival data of patients after medication will be collected and compared with the data of CONCEPT study, and multi-factor stratified analysis of the efficacy of voronib will be conducted.

DETAILED DESCRIPTION:
This is a multicenter real world study (RWS) initiated by the investigator. Eligible patients will be selected for treatment with second-line treatment including vorolanib and followed up. The real survival data of patients after medication will be collected and compared with the data of CONCEPT study, and multi-factor stratified analysis of the efficacy of voronib will be conducted. Vorolanib is a new generation of multi-target kinase inhibitors with a new chemical structure, which can inhibit tumor angiogenesis and growth, and is used in the treatment of various cancers. This multicenter, single-arm, open-labelled observational study is designed to include patients who meet the requirements for using vorolanib as a second-line treatment for renal cell carcinoma. For those patients who have reached the end point of the study, survival data during treatment with vorolanib is obtained for retrospective analysis. The patients who are still on treatment with vorolanib are followed up closely and survival data is obtained for prospective analysis. After summarizing the results of retrospective and prospective studies, relevant efficacy and safety conclusions will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have fully understood and voluntarily signed the informed consent form (ICF);
* 18-80 years old (at the time of signing the informed consent); Both men and women; ECOG PS score: 0-1;
* Renal cell carcinoma with clear cell components confirmed histologically or cytopathologically, including unresectable or recurrent metastatic renal cell carcinoma dominated by clear cell components;
* According to RECIST (version 1.1), there are targets that are considered to be observable;
* The main organs function well.

Exclusion Criteria:

* A history of malignancies other than the disease studied within the past 5 years, other than malignancies that are expected to be cured with treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery);
* Systemic treatment with other antitumor agents, including targeted agents, immunotherapy agents and their combination regimens (eligible for inclusion after 5 half-lives), local antitumor therapy, or clinical investigational drug or device therapy within 4 weeks prior to the initial study;
* Had major surgery within 4 weeks prior to initial study dosing (as judged by the investigator) or was in recovery;
* A history of severe drug allergy, including but not limited to antibody drugs;
* Patients with contraindications for immunotherapy restart;
* A known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation may require long-term adrenal corticosteroid therapy. Patients with thyroid, suprarenal, or hypopituitarism that can be controlled by hormone replacement therapy alone, type 1 diabetes mellitus, and psoriasis or vitiligo that do not require systemic treatment are eligible to participate in this study;
* Toxicity did not resolve after previous antitumor therapy, i.e., regression to baseline, NCI-CTCAE 5.0 level 0-1 (except for alopecia), or levels specified in inclusion/exclusion criteria. Irreversible toxicity (e.g., hearing loss) that is not reasonably expected to be aggravated by the drug under study may be included in the study;
* Have central nervous system metastases and/or cancerous meningitis;
* Known history of clinically significant liver disease, including those infected with viral hepatitis activity;
* Patients with uncontrolled third space effusion requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc. (Patients with no need to drain effusion or no significant increase in effusion after 3 days of stopping drainage could be included);
* Patients with any severe and/or uncontrolled disease;
* Renal failure requires hemodialysis or peritoneal dialysis;
* Have or have a suspected active autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc.;
* History of live attenuated vaccine vaccination within 4 weeks prior to the initial study or expected live attenuated vaccine vaccination during the study period;
* Those who have a history of psychotropic drug abuse and cannot abstain or have a history of mental disorders;
* Other severe, acute, or chronic medical or psychiatric conditions or laboratory abnormalities, as determined by the investigator, that may increase the risks associated with study participation or that may interfere with the interpretation of the study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects clinically diagnosed with advanced unresectable or metastatic renal cell carcinoma. After receiving at least one systemic therapy (including TKIs or TKIs combined with ICIs, including but not limited to axitinib, sunitinib, sorafenib, pembrolizumab, etc.), subjects reach PD as assessed by RECIST v1.1 and switch to second-line treatment options including vorolanib.
Sampling Method: Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From enrollment to the end of treatment at 12 weeks.
Treatment Related Adverse Events (TRAEs) | From enrollment to up to 90 days after treatment at 12 weeks or reported.

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to the end of treatment at 12 weeks.
Objective Response Rate (ORR) | From enrollment to the end of treatment at 12 weeks.
Disease Control Rate (DCR) | From enrollment to the end of treatment at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiu Liu, M. D., Study Chair — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China